CLINICAL TRIAL: NCT02822144
Title: General Anesthesia Versus Sedation During Intra-arterial Treatment for Stroke
Acronym: GASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC15_8957; 2016-000795-25 (EudraCT Number)
Record Dates: First submitted 2016-06-27; First posted 2016-07-04 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: ischemic stroke; thrombectomy; anesthesia; sedation
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Etomidate; Succinylcholine; Propofol; Remifentanil; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- general anesthesia (Experimental): General anesthesia with etomidate, succinylcholine, propofol and remifentanil
  Interventions: Drug: Etomidate; Drug: Succinylcholine; Drug: Propofol; Drug: Remifentanil
- sedation (Experimental): Sedation with remifentanil and local anesthesia with lidocaine
  Interventions: Drug: Remifentanil; Drug: Lidocaine

INTERVENTIONS:
Drug: Etomidate
  Arms: general anesthesia
Drug: Succinylcholine
  Arms: general anesthesia
Drug: Propofol
  Arms: general anesthesia
Drug: Remifentanil
Drug: Lidocaine
  Arms: sedation

SUMMARY:
In France, the annual incidence rate of acute ischaemic stroke is around 150 000 patients, 65 % of whom keep long-term disability. Several multicentric randomized controlled trials have shown the benefit of a mechanical thrombectomy in the acute phase of ischaemic stroke on functional disability, compared to a medical treatment alone (thrombolysis).

The timeliness of revascularisation is an essential factor of good prognosis. This intra-arterial treatment, associated with thrombolysis if applicable, is the reference treatment of large-vessel occlusion. The stillness of the patient is required to control the safety of the recanalization. Currently, either a general anesthesia or a sedation can be performed.

Several studies have shown a trend to superiority of the sedation but none was conducted with a high level of proof methodology.

The aim of our multicentric randomized controlled trial is to compare sedation and general anesthesia during intra-arterial thrombectomy for an acute ischaemic stroke in the anterior cerebral circulation. The main outcome will be the efficacy on the functional neurological prognosis at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Body mass index < or equal to 35 kg/m² ,
* Indication for thrombectomy, after multidisciplinary consultation,
* Proximal artery occlusion in the anterior circulation (internal carotid artery, M1, M2,...), confirmed on imaging (angioscan or angio-MRI),
* Written informed consent of the patient or a close / trusted person when possible, or emergency procedure,
* Patient affiliated to or beneficiary of an health insurance

Non-inclusion Criteria:

* Comorbidity committing short-term prognosis,
* Hemodynamic instability,
* Pregnant woman,
* Contra-indication to sedation: pre-existing swallowing impairment; restless patient, not able to stay lying down; Glasgow score < 8,
* Contra-indication to general anesthesia,
* Intubated patient at inclusion,
* Additional intracerebral hemorrhage,
* Sign of occlusion in a different cerebral territory,
* Known contra-indication to succinylcholine: hypersensitivity, hyperkaliemia,
* Known contra-indication to one of the anesthesic agents,
* Patient participating in another clinical trial, possibly interfering with the study procedures,
* Patient in a known situation of deprivation of freedom, guardianship or curatorship.

Exclusion criteria:

* Patients with deprivation of freedom will be excluded as soon as the investigator will have knowledge of the situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Score on the modified Rankin scale | 3 months

SECONDARY OUTCOMES:
Recanalization delay | Day 1
  Delay between first symptoms and last angiography
Delay between patient's hospitalization and start of procedure | Day 1
  At the time of puncture
Quality of recanalization assessed with TICI (Thrombolysis in cerebral infarction) score | Day 1
  At the last angiography
NIHSS score | Day 1
NIHSS score | Day 7
Angiographic complications: number of patients wtih dissection, arterial rupture, thrombus in another territory | Day 1
Mortality | 3 months
Number of episodes of hypo- / hypertension | 24 hours after thrombectomy
Number of patients with noradrenaline administration during anesthesia | Day 1
Number of sedations converted to general anesthesia and reason | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Axelle MAURICE, MD, Principal Investigator — Rennes University Hospital
Locations (4):
- France (4):
  - Département d'anesthésie-réanimation - Hôpital de la Cavale Blanche, CHU de Brest, Brest
  - Service d'anesthésie-réanimation - Fondation A. de Rothschild, Paris
  - Fédération d'anesthésie-réanimation - Hôpital Pontchaillou, CHU de Rennes, Rennes
  - Service d'anesthésie-réanimation 1 - Hôpital Bretonneau, CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maurice A, Eugene F, Ronziere T, Devys JM, Taylor G, Subileau A, Huet O, Gherbi H, Laffon M, Esvan M, Laviolle B, Beloeil H; GASS (General Anesthesia versus Sedation for Acute Stroke Treatment) Study Group and the French Society of Anesthesiologists (SFAR) Research Network. General Anesthesia versus Sedation, Both with Hemodynamic Control, during Intraarterial Treatment for Stroke: The GASS Randomized Trial. Anesthesiology. 2022 Apr 1;136(4):567-576. doi: 10.1097/ALN.0000000000004142. PMID 35226737
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365
- [Derived] Maurice A, Ferre JC, Ronziere T, Devys JM, Subileau A, Laffon M, Laviolle B, Beloeil H; SFAR research network. GASS Trial study protocol: a multicentre, single-blind, randomised clinical trial comparing general anaesthesia and sedation during intra-arterial treatment for stroke. BMJ Open. 2019 Jun 1;9(5):e024249. doi: 10.1136/bmjopen-2018-024249. PMID 31154292